CLINICAL TRIAL: NCT02081794
Title: Tailoring Patient Education to Perceived Risk for Falls in Hospitalized Oncology Patients: A Pilot Study
Brief Title: Tailoring Patient Education to Perceived Risk for Falls in Hospitalized Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE18Z13; NCI-2014-00388 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 18Z13 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Tailored education intervention) (Experimental): Participants receive a tailored educational intervention on the risk of falls comprising one of four two-minute videos determined by which educational group the participant is placed in: high risk/high perception, high risk/low perception, low risk/high perception, or low risk/low perception. Participants also receive tailored printed educational information concerning hospital falls based on the participants' answers given on the Perceived Risk Survey and are tailored to the participants' perception of falls risk. Participants also complete an investigator-constructed satisfaction survey at 24 and 72 hours post-intervention.
  Interventions: Other: Tailored education intervention
- Arm II (standard fall care) (Active Comparator): Participants receive standard care by nurses comprising a falls risk assessment and verbal education and receive an educational instruction sheet on falls prevention.
  Interventions: Other: Standard fall care

INTERVENTIONS:
Other: Tailored education intervention — Receive 2 minute video-assisted intervention on the risk and prevention of falls with tailored hand-outs depending on participant answers about fall risks
  Arms: Arm I (Tailored education intervention)
Other: Standard fall care — Patient are given a generic handout on falling and receive standard care by nurses comprising of a fall risk assessment and verbal education
  Arms: Arm II (standard fall care)

SUMMARY:
This randomized pilot clinical trial studies tailored patient educational intervention or standard education in assessing perceived risk for falls in hospitalized oncology patients. A tailored patient educational intervention may be more beneficial than standard education in preventing patients from falling by increasing the patient's knowledge of the risk factors for falling routinely and then providing education in deficit areas. Making patients more aware of the risk factors for falling may lead to greater engagement in preventative activities.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of a tailored, nurse-delivered intervention, as compared to the control group, on perceived risk for falls in hospitalized hematology-oncology patients.

II. To evaluate the effect of a tailored, nurse-delivered intervention, as compared to the control group, on confidence to minimize falls in hospitalized hematology-oncology patients.

III. To evaluate the relationship between patients' perceived risk for falling and their willingness to call for assistance with ambulation.

SECONDARY OBJECTIVES:

I. To evaluate the relationship between patients' perceived risk for falls and nursing risk assessments when using the standard hospital assessment tool and the investigator-designed perceived risk survey.

II. To evaluate the relationship between a patients' perceived risk for falls and sustaining a fall.

III. To evaluate patient satisfaction with the intervention.

OUTLINE:

All participants complete the Perceived Risk Survey comprising the participants' perceived risk for falls, their confidence to prevent a fall, and their willingness to ask for assistance at baseline and at 24 and 72 hours (or at discharge if stay is less than 72 hours) post-intervention. Patients are then randomized to 1 of 2 arms.

ARM I: Participants receive tailored education comprising one of four two-minute videos determined by which educational group the participant is placed in: high risk/high perception, high risk/low perception, low risk/high perception, or low risk/low perception. Participants also receive printed education sheets based on the participants' answers given on the Perceived Risk Survey and are tailored to the participants' perception of falls risk.

ARM II: Participants receive a generic educational instruction sheet on falls prevention and receive standard care by nurses comprising a falls risk assessment and verbal education.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer
* Admitted to the third floor of Seidman Cancer Center (SCC)
* Cognitively intact (alert, oriented to self, place, and time, and able to participate in the intervention)
* Ability to speak, read, and comprehend English

Exclusion Criteria:

* Nonmalignant diagnosis
* Actively dying
* Patients with a physician order for bed rest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Perceived risk for falls grouped according to the nurses assessment of risk using the University Hospitals (UH) Falls Assessment Tool | Up to 8 weeks
  Changes in pre vs post survey for the High Risk/Low Perception group will be compared to all others using a paired McNemar's test for both those receiving the intervention and controls. Pre and post scores will be compared between those receiving the intervention and controls using chi square tests.
Confidence to minimize falls assessed using the UH Falls Assessment Tool and the investigator-constructed Perceived Risk Survey (Nurse version) | Up to 8 weeks
  Pre vs post survey changes will be compared in confidence group using a paired McNemar's test for both those receiving the intervention and controls. Pre and post scores will be compared between those receiving the intervention and controls using chi square tests.
Willingness to call for assistance | Up to 8 weeks
  An eight-point Likert scale will be used. Pre vs post survey changes in willingness group will be compared using a paired McNemars test. Relationship between Risk/Perception group status and Willingness group will be assessed using a chi-square test stratified by pre or post survey results for both those receiving the intervention and controls.

SECONDARY OUTCOMES:
Relationship between patients perceived risk for falls and nurses risk assessments | Up to 8 weeks
  Descriptive statistics will be used to compare scores self-perceived risks of falling with a nurse's assessment of a patient falling
Patient's satisfaction of the intervention using the final questions on the Perceived Risk Post-Survey | Up to 8 weeks
  Descriptive statistics will be used by the distribution of pre vs post perceived risk values.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Kuhlenschmidt, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Seidman Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States